CLINICAL TRIAL: NCT06401668
Title: Impact of a Community Health Worker Strategy on Produce Prescription Program Uptake Among People With Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000037606; 24FIM1264456 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-05-01; First posted 2024-05-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Eligible participants will include primary and specialty care patients who identify as Hispanic with T2D and low incomes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRx with the CHW strategy (Experimental): Participants in this group will have CHWs to offer participants personalized support by overcoming barriers and leveraging facilitators to PRx uptake.
  Interventions: Behavioral: Community health worker (CHW) strategy; Behavioral: PRx Program
- PRx without the CHW strategy (Active Comparator): Participants in this group will participate in the PRx without the use of CHWs
  Interventions: Behavioral: PRx Program

INTERVENTIONS:
Behavioral: Community health worker (CHW) strategy — CHWs will offer participants personalized support to assist in overcoming barriers and leveraging facilitators to PRx uptake. CHWs are trained lay members of the communities they serve. The CHW strategy is an evidence-based.
  Arms: PRx with the CHW strategy
Behavioral: PRx Program — The PRx Program provides free fruit and vegetables and nutrition education to patients with T2D and food insecurity.

SUMMARY:
Produce prescription programs (PRx) are promising interventions for improving health outcomes for patients with both type 2 diabetes (T2D) and food insecurity, but uptake has been suboptimal. There is a critical need for scalable, evidence-based implementation strategies for improving PRx uptake and optimizing the effectiveness and cost-effectiveness of these interventions. This study will co-design and pilot a community health worker (CHW) strategy and test the effectiveness of the strategy compared to PRx participants without a CHW. The overall objective of this study is to test and evaluate a theory-informed, user-centered community health worker (CHW) implementation strategy to improve uptake of a PRx, among Hispanic Medicaid-eligible patients with T2D in Connecticut (CT). CHWs will offer participants personalized support by overcoming barriers and leveraging facilitators to PRx uptake.

DETAILED DESCRIPTION:
This study will have a small pilot followed by a randomized controlled trial. The focus of this registration is the randomized controlled trial.

First, following community co-design of the CHW strategy, investigators will conduct a two-month pilot study with an anticipated 10 participants to test the CHW strategy, the produce prescription program Rx, and overall study procedures. All participants will receive the PRx program with CHW strategy for two months.

Second, a randomized controlled trial to evaluate the effectiveness of the CHW strategy on barriers to PRx uptake, level of PRx engagement, and short-term program, behavioral, and health outcomes will be conducted.

Investigators hypothesize that participants who receive added CHW support during their enrollment in the PRx program will have reduced barriers to PRx uptake, higher PRx uptake, and greater improvements in the defined short-term program outcomes compared with participants who do not receive the CHW support during their enrollment in the PRx.

ELIGIBILITY:
Inclusion Criteria:

* Be a current primary or specialty care patient at Hartford Hospital
* Live in Hartford County
* Identify as Hispanic
* Have a current diagnosis of Type II Diabetes
* Be eligible for Medicaid based on household income and size.

Exclusion Criteria:

* Does not speak English or Spanish
* Has a diagnosis of gestational diabetes
* Individuals who are members of vulnerable populations, such as individuals who are incarcerated and individuals who are not able to consent.

Participants who are pregnant will be eligible for the study if they meet all of the inclusion criteria and do not have any of the exclusion criteria, as the study activities (additional funds to purchase fruits and vegetables, nutrition education, and support from a Community Health Worker) does not pose any additional risk to this group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PRx redemption | Monthly, beginning 1 month after the study start though the end of the six month study period.
  PRx redemption is defined as produce debit card dollars used/total dollars available will be collected from the produce debit card platform.

SECONDARY OUTCOMES:
Barriers to PRx uptake | 3 months, 6 months
  Barriers to PRx uptake will be captured through post-program survey questions on participant barriers to buying and consuming produce as well as from listening sessions and CHW process tracking data on participant encounters.
PRx uptake: Initiation | 6 months
  PRx initiation defined as the number of participants initiating use of the debit card/number enrolled
PRx uptake: Usage | 6 months
  • Months used (defined as #/% participants using any incentives each month for 6mo and % using incentives every month)
PRx uptake: Attendance | 6 months
  Nutrition class attendance defined as a yes/no variable for each of the three classes.
Program Satisfaction | 6 months
  Assessed through listening sessions and a short satisfaction module, coded on a five-point Likert scale in the post survey. Total score range from 0-4 with higher scores indicating greater satisfaction.
Change in Fruit and Vegetable Intake | baseline, 3 months, and 6 months
  Assessed with the 29-item Diet Quality Questionnaire. The 5-minute module asks yes/no questions about consumption of a series of sentinel foods that correspond to pre-defined food groups. It has a total score of 0-10. The higher the score, the higher the likelihood of nutrient adequacy.
Change in Household Food Insecurity | baseline, 3 months, and 6 months
  Assessed using the 6-item US Department of Agriculture Household Food Security Survey Module. The total score range from 0 to 27, with higher scores indicating more food security.
Change in Glycemic control | baseline and 6 months
  Assessed with HbA1c concentration (%) data from patient electronic medical records. A decrease in HbA1c concentration indicates better glycemic control.
Change in Self-rated Health | baseline, 3 months, and 6 months
  Assessed with a single question with a five-item response scale from poor to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perez-Escamilla, MD, Principal Investigator — Yale School of Public Health
Locations (1):
- Hartford HealthCare/ St. Vincent Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated within this study will be provided to the American Heart Association in a de-identified form, to be deposited within the Health Care x Food data repository on the Precision Medicine Platform, and subject to the Precision Medicine Platform Terms and Conditions. Data on the Precision Medicine Platform will be collated with data from other studies that are funded by the American Heart Association Health Care x Food initiative, and used by future investigators for analysis. In addition, data will be made available on Clinicaltrials.gov in alignment with agreed-upon Open Science Policies at the American Heart Association, whereby any factual data that is needed for independent verification of research results must be made freely and publicly available in an AHA-approved repository as soon as possible, and no later than the time of an associated publication or the end of the award period (and any no-cost extension), whichever come first.